CLINICAL TRIAL: NCT05409144
Title: Impact of Thoracic Epidural Infusion Versus Continuous Serratus Anterior Plane Block Versus Continuous Erector Spinae Plane Block on Incidence of Post Thoracotomy Pain Syndrome: A Randomized Controlled Trial
Brief Title: Impact of Thoracic Epidural Versus Serratus Anterior Plane Block Versus Erector Spinae Plane Block on Incidence of PTPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Shaban Mohammed, assisstant lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2202-30106
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Post-thoracotomy Pain Syndrome; Erector Spinae Plane Block; Serratus Anterior Plane Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic epidural infusion group (Experimental): Patients will receive thoracic epidural preoperative
  Interventions: Procedure: Thoracic epidural infusion
- Erector Spinae Plane Block group (Experimental): Patients will receive Ultrasound-guided Erector Spinae Plane Block preoperative with an injection of 30 ml levobupivacaine 0.25% and insertion of a catheter
  Interventions: Device: Erector Spinae Plane Block
- Serratus Anterior Plane Block group (Experimental): Patients will receive Ultrasound-guided Serratus Anterior Plane Block preoperative with an injection of 30 ml levobupivacaine 0.25%.
  Interventions: Device: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Thoracic epidural infusion — Upon locating the desired site spot, lidocaine 1% must be injected into the skin and underlying tissues to decrease the discomfort with the advancement of the epidural needle. Once achieving local anesthesia, the epidural needle advanced with its stylet in place and with its bevel point cephalad; this will ultimately contribute to the proper location of the epidural catheter. The epidural needle must be advanced through the skin, subcutaneous tissue, supraspinous, and interspinous ligaments. Once there, the stylet must be removed, and the Loss of Resistance syringe (filled up with saline, air, or both) must be attached to the needle. The needle must be advanced while applying pressure to the plunger. Once the ligamentum flavum is pierced, a loss in resistance will be noted; this is the epidural space, and 5 to 10 cc of saline is injected to expand the epidural space; this may decrease the risk of vascular injury.
  Arms: Thoracic epidural infusion group
Device: Erector Spinae Plane Block — The block-level will be at T5. The ultrasound probe will be placed on the back in a transverse orientation to identify the tip of the T5 transverse process; these are recognizable as flat, squared-off acoustic shadows with only a very faint image of the pleura visible. The tip of the transverse process will be centered on the ultrasound screen and the probe will then be rotated into a longitudinal orientation to produce a parasagittal view, in which the following layers will be visible superficial to the acoustic shadows of the transverse processes: skin and subcutaneous tissue, trapezius, erector spinae muscle and T5 transverse process. 3ml lidocaine 1% will be used on skin and subcutaneous fat, Echogenic block needle will be inserted in-plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T5 transverse process.
  Arms: Erector Spinae Plane Block group
Device: Serratus Anterior Plane Block — The block is performed with full aseptic precautions. Arm abduction is preferred. The ultrasound probe will be placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib, with the indicator oriented toward the operator's left. With the rib, pleural line, and overlying serratus anterior and latissimus dorsi muscles visualized, then, 3ml lidocaine 1% will be used for skin and subcutaneous fat, using ultrasound guidance, a 38-mm 22-gauge regional block needle is going to be advanced in-plane at an angle of approximately 45 degrees towards the fifth rib. After aspiration to avoid intravascular injection 30ml of levobupivacaine 0.25% will be injected anteriorly to the rib and deep into the serratus anterior muscle.
  Arms: Serratus Anterior Plane Block group

SUMMARY:
The aim of this study is to evaluate the impact of Ultrasound-guided Erector Spinae plane block compared to Ultrasound-guided serratus anterior plane block on the emergence of post-thoracotomy pain syndrome in patients undergoing lobectomy for lung cancer.

DETAILED DESCRIPTION:
Lung cancer has the highest incidence of all malignancies worldwide and accounts for approximately 13% of all cancer cases. Lung cancer is still the most common cause of cancer-related deaths, and lung resection surgeries could be the main therapeutic option. Hence, the number of thoracotomy procedures is progressively increasing as is the incidence of post-thoracotomy pain. In addition to amputation and mastectomy, thoracotomy is considered the main etiology of severe and long-term acute and chronic post-surgical pain syndromes (CPSPs). The prevalence of post-thoracotomy pain syndrome (PTPS) is widely variable (30%-50%) and may range from 11% to 80%, according to other studies.

The International Association for the Study of Pain (IASP) has defined post-thoracotomy pain syndrome as "pain that recurs or persists along the thoracotomy scar at least 2 months after the procedure". In addition, post-thoracotomy pain syndrome is mostly described with neuropathic manifestations along the thoracotomy scar and in the mammary, inframammary, ipsilateral scapular and interscapular areas.

The ultrasound-guided erector spinae plane (ESP) block is a novel technique for thoracic analgesia that promises to be a relatively simple and safe alternative to more complex and invasive techniques of neural blockade.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-65) Years
* Physical status American Society of Anesthesiologists Classification II, III
* Patients undergoing lobectomy through lateral thoracotomy
* Body mass index (BMI): (20-40) kg/m2

Exclusion Criteria:

* Patient refusal.
* Age <18 years or >65 years
* Body mass index (BMI) <20 kg/m2 and >40 kg/m2
* Known sensitivity or contraindication to drugs used in the study
* Contraindication to regional anesthesia e.g. local infection at site of introduction, pre-existing peripheral neuropathies and coagulopathy.
* Pregnancy.
* Physical status American Society of Anesthesiologists Classification IV
* patients on chronic analgesic therapy (daily morphine ≥30 mg or equivalent dose of other opioids or tramadol or any medication for neuropathic pain)
* patients with a history of drug abuse
* patients with neuropsychiatric diseases; patients with a history of chronic pain syndromes that may enhance sensitivity to pain, for example, fibromyalgia
* patients with a history of thoracic surgery through lateral thoracotomy; and patients with recurrent chest malignancies within 3 months.
* All patients who developed severe intra- or post-operative bleeding or required postoperative mechanical ventilation were also excluded from the study.
* Thoracic spine disorders or deformity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients developing post-thoracotomy pain syndrome | 12 weeks postoperatively
  The incidence of patients developing post-thoracotomy pain syndrome according to grading system for neuropathic pain (GSNP

SECONDARY OUTCOMES:
Morphine consumption | 48 hours Postoperatively
  The total amount of morphine consumed postoperatively for 48 hours.
Fentanyl consumption | Intraoperatively
  Total amount of fentanyl consumed intraoperative
Post-thoracotomy pain syndrome severity | 12 weeks postoperatively
  Severity of Post-thoracotomy pain syndrome according to Grading system for neuropathic pain (GSNP)
Patient's Quality of life | 12 weeks postoperatively
  Patient's Quality of life according to the Flanagan Quality of Life Scale (QOLS)
Postoperative Patient's activity level | 12 weeks postoperatively
  Postoperative Patient's activity level according to Barthel Activities of Daily Living scale (ADL)
Heart rate | Intraoperatively
  Heart rate will be recorded
Mean arterial blood pressure | Intraoperatively
  Mean arterial blood pressure will be recorded
Nausea and vomiting | 24 hours postopertivley
  Postoperative nausea and vomiting (PONV) will be recorded
Post-operative pain | 24 hours postopratively
  Post-operative pain will be assessed by the Numeric Rating Scale (NRS)
Time taken till 1st rescue analgesic request | 24 hours postopratively
  The time till administration of first rescue analgesia will be recorded
Postoperative pulmonary complications | 24 hours postopratively
  Postoperative pulmonary complications will be recorded

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the author
Supporting Information: Study Protocol
Time Frame: One year after the study is ended